CLINICAL TRIAL: NCT03604224
Title: Retrospective Observational Study to Observe Clinical Effectiveness of Canagliflozin 300 mg Containing Treatment Regimens in Indian Type 2 Diabetes Patients With BMI>25 kg/m^2, in Real World Clinical Setting
Brief Title: A Study to Observe Clinical Effectiveness of Canagliflozin 300 mg Containing Treatment Regimens in Indian Type 2 Diabetes Participants With BMI>25 kg/m^2, in Real World Clinical Setting
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108507; 28431754DIA4030 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Canagliflozin Containing Treatment Regimens: No intervention will be administered as a part of this study. Participants with type 2 diabetes mellitus (T2DM) who were initiated on canagliflozin 300 milligram (mg) treatment 12 weeks back and meeting the inclusion criteria will be observed.
  Interventions: Drug: Canagliflozin 300 mg

INTERVENTIONS:
Drug: Canagliflozin 300 mg — Participants who are initiated on canagliflozin 300 mg will be observed. No study treatment will be administered as a part of this study.

SUMMARY:
The purpose of this study is to observe clinical effectiveness of canagliflozin by mean haemoglobin A1c (HbA1C) and body weight changes from baseline to 12 weeks in Indian type 2 diabetes participants.

ELIGIBILITY:
Inclusion Criteria:

* T2DM participants on a stable anti-hyperglycemic regimen containing one or more anti-diabetic drug for at least 30 days and had HbA1c of more than 7 percent (%) at the time of, or within 2 weeks before canagliflozin 300 mg initiation
* T2DM participants as confirmed from hospital records
* T2DM participant having BMI>25kg/m^2 at the time of canagliflozin 300 mg initiation
* Participants having clinical assessment data (at least glycated haemoglobin A1c [HbA1c] and body weight) for at least two visits, that is (i.e.) visit at which treatment with canagliflozin 300 mg was initiated or 2 weeks before initiation and follow-up visit at 12 weeks (+-4 weeks) from initiation, in accordance with the usual clinical practice

Exclusion Criteria:

* Participants with history of autoimmune diabetes (type 1 diabetes mellitus [T1DM] or latent autoimmune diabetes in adults [LADA]), pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy or gestational diabetes or any off-label use or patient data refusal based on physician discretion
* Participants with a history of use of other Sodium Glucose co-Transporter 2 (SGLT2) inhibitor within 12 weeks (empagliflozin or dapagliflozin)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include Indian type 2 diabetes mellitus (T2DM) participants with body mass index (BMI) greater than (>)25 kilogram per meter square (kg/m^2), initiated canagliflozin 300 milligram (mg) as part of their treatment regimens, in real world clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Mean Hemoglobin A1c (HbA1c) | Baseline up to 12 weeks
  Change in mean HbA1c from baseline to 12 weeks will be determined. HbA1c refers to glycated haemoglobin (A1c), which identifies average plasma glucose concentration.
Change From Baseline in Mean Weight | Baseline up to 12 weeks
  Change in mean body weight from baseline to 12 weeks will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (3):
- India (3):
  - Diacon Hospital, Bangalore
  - Dr. A. Ramachandran's Diabetes Hospitals, Chennai
  - Apollo Hospitals, Kolkata